CLINICAL TRIAL: NCT01124188
Title: Optimizing Care for Older Adults With Back Pain and Depression
Brief Title: ADAPT: Addressing Depression and Pain Together
Acronym: ADAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jordan F. Karp, Associate Professor of Psychiatry, Anesthesiology, and Clinical and Translational Science, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG033575
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Depression; Back Pain
Keywords: Geriatric psychiatry; Aged; Elderly; Venlafaxine; Self efficacy; Pain; Psychotherapy; Effexor
MeSH Terms: conditions — Depression; Back Pain; Pain | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Intervention Arm (Experimental): Higher-dose venlafaxine and Problem Solving Therapy for Depression and Pain (PST-DP)
  Interventions: Drug: Higher-dose venlafaxine; Behavioral: Problem Solving Therapy for Depression and Pain
- Active Control (Active Comparator): Higher-dose venlafaxine and supportive management (SM)
  Interventions: Drug: Higher-dose venlafaxine; Behavioral: Supportive management

INTERVENTIONS:
Drug: Higher-dose venlafaxine — Dosing of venlafaxine will range from 187.5-300 mg/day.
  Other Names: Effexor
Behavioral: Supportive management — Supportive management encourages participants to take the medication and manages any treatment-emergent side effects. Ten sessions will be delivered over the course of 14 weeks.
  Arms: Active Control
Behavioral: Problem Solving Therapy for Depression and Pain — PST-DP will be delivered over the course of 10 sessions over 14 weeks. Along with teaching the participant 7 steps of problem solving, PST-DP also includes a medication support and management component.
  Other Names: PST-DP
  Arms: Study Intervention Arm

SUMMARY:
The primary question addressed by this study is: Using a stepped care approach in primary care, what is the value of the combination of an antidepressant medication (Venlafaxine) and psychotherapy for seniors living with depression and chronic lower back pain when treatment with a low-dose of venlafaxine and supportive management (SM) has led to only a partial or non-response?

DETAILED DESCRIPTION:
The primary aims of the study are:

1. To test the efficacy of higher-dose Venlafaxine and Problem Solving Therapy for Depression and Pain (VEN/PST-DP) in reducing depression and pain.
2. To test the efficacy of higher-dose VEN/PST-DP in reducing back-related disability and improving physical functioning.

Primary Hypotheses:

1. During the 14 weeks of step 2, patients receiving VEN/PST-DP, compared to those receiving VEN/SM, will respond faster and have a higher rate of response.
2. During the 14 weeks of phase 2, patients receiving VEN/PST-DP, compared to those receiving VEN/SM, will have better self-reported physical functioning.

   Secondary Hypothesis:
3. Self-efficacy has been shown to predict treatment outcomes for both depression and pain. We have observed that the self-efficacy for pain management of these patients improves with antidepressant pharmacotherapy. We hypothesize that for subjects assigned to receive treatment with VEN/PST-DP, self-efficacy will mediate treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 or older
2. Scores 10 or higher on the Patient Health Questionnaire-9 (PHQ-9). This is consistent with at least moderate depression severity.
3. Endorses low back pain more days than not, of at least moderate severity, for at least the past 3 months.
4. If venlafaxine up to 150 mg/day has been tried for at least 6 weeks, subjects must have been *completely* unresponsive for both depression and low back pain (based on subject report).
5. During this episode of CLBP, must have tried without continued success any of the following: 1) prescription or over the counter analgesics, 2) physical therapy, 3) acupuncture, 4) injection therapy, 5) had back surgery, 6) multidisciplinary pain program, 7) psychological treatment for chronic pain such as cognitive behavioral therapy or biofeedback, or 8) any other physician-prescribed treatment for chronic low back pain.

Upon meeting, after obtaining written informed consent, the following inclusion criteria are administered to determine protocol-eligibility:

1. Repeat PHQ-9 with score
2. Current depression (major depression, partial remission of major depression, minor depression, or dysthymia) diagnosed with the PRIMEMD
3. 20-item Numeric Rating Scale for low back pain
4. The Montreal Cognitive Assessment (MoCA). Eligibility requires score of at least 24
5. No history of alcohol/substance abuse or dependence for the past six months. If subjects took more analgesics than prescribed for CLBP but there was no other evidence of abuse, they will be included. Alcohol and substance abuse will be assessed with the MINI-International Neuropsychiatric Interview.

Exclusion Criteria:

The following exclusion criteria will be assessed during telephone screening. If the individual responds in the affirmative to any of these conditions, they will not be eligible:

1. Wheelchair-bound as this level of disability does not represent most older adults living with CLBP.
2. Diagnosed with fibromyalgia; there is evidence that individuals with fibromyalgia may have a differential treatment response to SNRIs.
3. Involved in a lawsuit related to back pain and/or receiving workers compensation.

Subjects must also not meet any of the following exclusion criteria:

1. Current or past psychotic-spectrum disorder or current or past bipolar disorder. This will be determined with the PRIME-MD and MINI-Neuropsychiatric interview.
2. Medically unstable, delirious, or terminally ill; or medical contraindication to use of venlafaxine therapy, including hypersensitivity, history of venlafaxine-induced SIADH, uncontrolled narrow angle glaucoma, AST or ALT > 1.5x upper limit of normal.
3. Acute low back pain "red flag" superimposed on chronic low back pain suggesting medically emergent condition (e.g., vertebral fracture, infection, cauda equina syndrome, disk herniation, cancer).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan F Karp, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Late Life Depression Program, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karp JF, Weiner DK, Dew MA, Begley A, Miller MD, Reynolds CF 3rd. Duloxetine and care management treatment of older adults with comorbid major depressive disorder and chronic low back pain: results of an open-label pilot study. Int J Geriatr Psychiatry. 2010 Jun;25(6):633-42. doi: 10.1002/gps.2386. PMID 19750557
- [Background] Karp JF, Skidmore E, Lotz M, Lenze E, Dew MA, Reynolds CF 3rd. Use of the late-life function and disability instrument to assess disability in major depression. J Am Geriatr Soc. 2009 Sep;57(9):1612-9. doi: 10.1111/j.1532-5415.2009.02398.x. Epub 2009 Jul 21. PMID 19682111
- [Background] Karp JF, Reynolds CF 3rd, Butters MA, Dew MA, Mazumdar S, Begley AE, Lenze E, Weiner DK. The relationship between pain and mental flexibility in older adult pain clinic patients. Pain Med. 2006 Sep-Oct;7(5):444-52. doi: 10.1111/j.1526-4637.2006.00212.x. PMID 17014605
- [Background] Karp JF, Weiner D, Seligman K, Butters M, Miller M, Frank E, Stack J, Mulsant BH, Pollock B, Dew MA, Kupfer DJ, Reynolds CF 3rd. Body pain and treatment response in late-life depression. Am J Geriatr Psychiatry. 2005 Mar;13(3):188-94. doi: 10.1176/appi.ajgp.13.3.188. PMID 15728749
- [Background] Arean P, Hegel M, Vannoy S, Fan MY, Unuzter J. Effectiveness of problem-solving therapy for older, primary care patients with depression: results from the IMPACT project. Gerontologist. 2008 Jun;48(3):311-23. doi: 10.1093/geront/48.3.311. PMID 18591356
- [Background] Karp JF, Shega JW, Morone NE, Weiner DK. Advances in understanding the mechanisms and management of persistent pain in older adults. Br J Anaesth. 2008 Jul;101(1):111-20. doi: 10.1093/bja/aen090. Epub 2008 May 16. PMID 18487247
- [Derived] Stahl ST, Jung C, Weiner DK, Pecina M, Karp JF. Opioid Exposure Negatively Affects Antidepressant Response to Venlafaxine in Older Adults with Chronic Low Back Pain and Depression. Pain Med. 2020 Aug 1;21(8):1538-1545. doi: 10.1093/pm/pnz279. PMID 31633789
- [Derived] Wei W, Karim HT, Lin C, Mizuno A, Andreescu C, Karp JF, Reynolds CF 3rd, Aizenstein HJ. Trajectories in Cerebral Blood Flow Following Antidepressant Treatment in Late-Life Depression: Support for the Vascular Depression Hypothesis. J Clin Psychiatry. 2018 Oct 23;79(6):18m12106. doi: 10.4088/JCP.18m12106. PMID 30358242
- [Derived] Rej S, Dew MA, Karp JF. Treating concurrent chronic low back pain and depression with low-dose venlafaxine: an initial identification of "easy-to-use" clinical predictors of early response. Pain Med. 2014 Jul;15(7):1154-62. doi: 10.1111/pme.12456. Epub 2014 Jul 4. PMID 25040462
- See also: The Late-Life Depression Evaluation and Treatment Center provides information and treatment for depression, anxiety disorders, and insomnia in older Americans. — http://www.wpic.pitt.edu/research/
- See also: The University of Pittsburgh Institute on Aging provides access to a multidisciplinary network of comprehensive clinical care. — http://www.aging.pitt.edu/
- See also: The American Association for Geriatric Psychiatry is a national association representing and serving its members and the field of geriatric psychiatry. — http://www.aagpgpa.org/
- See also: website describing the study — http://www.ADAPTstudy.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Intervention Arm: Higher-dose venlafaxine and Problem Solving Therapy for Depression and Pain (PST-DP)
  Combination Treatment with Higher-dose venlafaxine + PST-DP: Dosing of venlafaxine will range from 187.5-300 mg/day. Medication management and PST-DP will be delivered over the course of 10 sessions over 14 weeks.
- Active Control: Higher-dose venlafaxine and supportive management (SM)
  Higher-dose venlafaxine and supportive management: The dose of venlafaxine will be between 187.5-300 mg/day. It will be offered with supportive management which encourages participants to take the medication and manages any treatment-emergent side effects. Ten sessions will be delivered over the course of 14 weeks.
Period: Overall Study
Arm/Group | Study Intervention Arm | Active Control
Started | 68 | 71
Completed | 60 | 65
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Intervention Arm | Active Control | Total
Number analyzed (Participants) | 68 | 71 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 33 | 50
  >=65 years | 51 | 38 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.81 (7.90) | 69.90 (8.73) | 70.34 (8.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 27 | 26 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68 | 71 | 139

OUTCOME MEASURES:

1. Primary Outcome: Proportion Responding Initially by Treatment Arm During 14 Weeks Post Randomization
Description: The PHQ-9 depression questionnaire scores range from 0 to 27. The higher the score the more severe the depression. A PHQ-9 score less than or equal to 5 represents absence of depression. The Numeric Rating scale is a self report pain scale ranging from 0 to 20. Higher numbers indicate more pain. Response in this study was defined as two consecutive PHQ-9 scores < or = to 5 AND Numeric Rating Scale for pain (NRS) > or = 30% reduction from study entry.
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Study Intervention Arm | Active Control
Number analyzed (Participants) | 68 | 71
Participants | 28 | 28
Statistical Analysis 1: Comparison: Study Intervention Arm vs Active Control; Test type: Superiority or Other; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.63 to 1.80]

2. Secondary Outcome: Change in Roland Morris Disability Questionnaire (RMDQ) From P2 Baseline to 14 Weeks
Description: Change in RMDQ from randomization to 14 weeks. The Roland-Morris is a 24-item self-report questionnaire about how low-back pain affects functional activities. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability).
  Improvement of 30% is clinically meaningful
Time Frame: Baseline and 14 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Study Intervention Arm | Active Control
Number analyzed (Participants) | 68 | 71
units on a scale | -3.67 [-4.88 to -2.46] | -3.20 [-4.35 to -2.05]
Statistical Analysis 1: Comparison: Study Intervention Arm vs Active Control; Test type: Superiority or Other; p = .49, Mixed Models Analysis

3. Secondary Outcome: Changes in Short Physical Performance Battery From Ph 2 Baseline Till 14 Weeks
Description: Change in SPPB scores from randomization to 14 weeks for both arms.
  The Short Physical Performance Battery (SPPB) assesses physical performance. The SPPB scores range from 0-12 and assess lower extremity strength, balance, and gait speed, three meaningful predictors of morbidity and mortality in late-life. Lower scores on the SPPB indicates greater limitations. Improvement of 0.5 points indicate clinically meaningful improvement in physical performance
Time Frame: Baseline and 14 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Study Intervention Arm | Active Control
Number analyzed (Participants) | 68 | 71
units on a scale | 0.49 [-0.06 to 1.03] | 0.54 [0.06 to 1.02]
Statistical Analysis 1: Comparison: Study Intervention Arm vs Active Control; Test type: Superiority or Other; p = 0.88, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Study Intervention Arm | Active Control
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No